CLINICAL TRIAL: NCT05630547
Title: A Phase 2 Double-blind, Randomized, Placebo-controlled Study Evaluating the Effect of SAR443820 on Serum Neurofilament Levels in Participants With Multiple Sclerosis, Followed by an Open-label Long-term Extension Period
Brief Title: A Study to Evaluate the Effect of SAR443820 on Serum Neurofilament Levels in Male and Female Adult Participants With Multiple Sclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated as it did not meet its primary and key secondary endpoints
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT16753; U1111-1271-1257 (Registry Identifier: ICTRP); ACT16753 (Other: Sanofi Identifier); 2023-509078-45-00 (Registry Identifier: CTIS); 2022-000049-34 (EudraCT Number)
Record Dates: First submitted 2022-11-07; First posted 2022-11-29 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded treatment (Part A) and open-label long-term extension period (Part B)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAR443820 (Experimental): Oral SAR443820
  Interventions: Drug: SAR443820
- Placebo (Placebo Comparator): Oral placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SAR443820 — Tablet by oral administration
  Arms: SAR443820
Other: Placebo — Tablet by oral administration
  Arms: Placebo

SUMMARY:
This was a Phase 2, randomized, double-blind, placebo-controlled 2 parallel-arm study to assess the effect on serum neurofilament light chain (sNfL), safety and tolerability of oral SAR443820 compared to placebo in male and female participants aged 18 to 60 years with relapsing-remitting multiple sclerosis (RRMS), secondary progressive multiple sclerosis (SPMS) (relapsing or non-relapsing), or primary progressive multiple sclerosis (PPMS) followed by an open-label long-term extension period.

The total study duration was approximately 100 weeks and included the following:

4-week screening period 48-week double-blind treatment period (Part A) 48-week open-label long-term extension period (Part B)

The study was terminated prior to completion (of Week 96) as primary endpoint was not met. Therefore final duration was less than 96 weeks.

DETAILED DESCRIPTION:
Approximately 100 weeks

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 60 years (inclusive) of age, at the time of signing the informed consent.
* Participants with diagnosis of RRMS, SPMS (relapsing or non-relapsing) or primary progressive subtype according to the 2017 revision of the McDonald diagnostic criteria (SPMS diagnostic criteria according to initial relapsing remitting disease course followed by progression with or without occasional relapses, minor remissions, and plateaus; progression denotes the continuous worsening of neurological impairment over at least 6 months).
* Participants with Expanded Disability Status Scale (EDSS) score of 2 to 6 inclusive at screening.
* Participants who were either untreated or in the opinion of the Investigator were stable on an allowed disease-modifying therapy (DMT) (interferons, glatiramer acetate, fumarates, or teriflunomide) for at least the past 3 months, AND not anticipated to require a change in multiple sclerosis (MS) treatment for the duration of Part A and Part B (through Week 96); in Part B changes in dose of allowed DMTs or transition to other allowed DMTs was permitted).
* Participants with body weight at least 45 kg and body mass index (BMI) at least 18.0 kg/m^2.
* Contraceptive use by men and women was consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Participants with immunodeficiency syndromes or other autoimmune diseases requiring immunosuppressive therapy
* Participants with a history of seizures or epilepsy (history of febrile seizure during childhood was allowed).
* Participants with known clinical relapse (acute or subacute episodes of new or increasing neurological dysfunction followed by full or partial recovery, in absence of fever or infection) within 8 weeks of screening.
* Participants with neurological disease history other than MS, eg, head trauma within 3 months, cerebrovascular disease, and vascular dementia.
* Participants with a history of recent serious infection (eg, pneumonia, septicemia) within 4 weeks of screening; an infection requiring hospitalization or intravenous antibiotics, antivirals, or antifungals within 4 weeks of screening; or chronic bacterial infections (such as tuberculosis) deemed unacceptable, as per Investigator's judgment.
* Participants who had significant cognitive impairment, psychiatric disease, other neurodegenerative disorders (eg, Parkinson disease or Alzheimer disease), substance abuse, or any other conditions that made the participants unsuitable for participating in the study or interfered with assessment or completing the study in the opinion of the Investigator.
* Participants with a documented history of attempted suicide over the 24 weeks prior to the Screening Visit, presents with suicidal ideation of category 4 or 5 on the Columbia Suicide Severity Rating Scale (CSSRS), or if in the Investigator's judgment, the participant was at risk for a suicide attempt.
* Participants with a history of unstable or severe cardiac, pulmonary, oncological, hepatic, or renal disease or another medically significant illness other than MS precluding their safe participation in this study.
* Participants who received a live vaccine within 14 days before the Screening Visit.
* Participants with a known history of allergy to any ingredients of SAR443820 (mannitol, lactose monohydrate, sodium starch glycolate, colloidal silicon dioxide, magnesium stearate, hypromellose, titanium dioxide, polyethylene glycol, and microcrystalline cellulose).
* Participants who used any medications that are moderate or strong inhibitors or strong inducers of cytochrome P450 3A4 (CYP3A4).
* Participants who used of any of the following medications/treatments: fampridine/dalfampridine, ofatumumab, fingolimod, cladribine, siponimod, ponesimod, ozanimod, alemtuzumab, mitoxantrone, ocrelizumab, natalizumab, or similar approved compounds but with different trade names and any unapproved treatments or therapies for MS; any DMTs newly approved after January 2023 that are marketed at any time during the course of the double-blind study period. These medications were not allowed within 5 half-lives before the Screening Visit and for the duration of Part A and Part B.
* Participants who had prior/concurrent clinical study enrollment, ie, the participant had taken other investigational drugs within 4 weeks or 5 half-lives, whichever was longer, before the first Screening Visit; concurrent or recent participation in non-interventional studies may be permitted.

Participants with abnormal laboratory test(s) at the Screening Visit:

* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) more than 3.0 x upper limit of normal (ULN)
* Bilirubin more than 1.5 x ULN; unless the participant has documented Gilbert syndrome (isolated bilirubin more than 1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%)
* Serum albumin less than 3.5 g/dL
* Estimated Glomerular filtration rate less than 60 mL/min/1.73 m^2 (Modification of Diet in Renal Disease [MDRD])
* Other abnormal laboratory values or electrocardiogram (ECG) changes that are deemed clinically significant as per Investigator's judgment
* The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (35):
- Belgium (3):
  - Investigational Site Number : 0560001, Brussels
  - Investigational Site Number : 0560002, Ghent
  - Investigational Site Number : 0560003, Overpelt
- Bulgaria (3):
  - Investigational Site Number : 1000001, Sofia
  - Investigational Site Number : 1000002, Sofia
  - Investigational Site Number : 1000003, Sofia
- Canada (4):
  - Investigational Site Number : 1240002, Ottawa, Ontario
  - Investigational Site Number : 1240004, Toronto, Ontario
  - Investigational Site Number : 1240001, Gatineau, Quebec
  - Investigational Site Number : 1240003, Lévis, Quebec
- Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago, Chile
- China (4):
  - Investigational Site Number : 1560003, Chengdu
  - Investigational Site Number : 1560002, Shanghai
  - Investigational Site Number : 1560001, Tianjin
  - Investigational Site Number : 1560004, Xi'an
- France (4):
  - Investigational Site Number : 2500004, Caen
  - Investigational Site Number : 2500002, Nice
  - Investigational Site Number : 2500001, Paris
  - Investigational Site Number : 2500003, Strasbourg
- Investigational Site Number : 2760002, Würzburg, Germany
- Italy (4):
  - Investigational Site Number : 3800001, Pozzilli, Isernia
  - Investigational Site Number : 3800005, Cagliari
  - Investigational Site Number : 3800002, Milan
  - Investigational Site Number : 3800003, Milan
- Poland (5):
  - Investigational Site Number : 6160004, Plewiska, Greater Poland Voivodeship
  - Investigational Site Number : 6160002, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160005, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160001, Krakow
  - Investigational Site Number : 6160006, Zabrze
- Spain (6):
  - Investigational Site Number : 7240002, Seville, Andalusia
  - Investigational Site Number : 7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240003, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240004, Madrid / Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240006, Madrid
  - Investigational Site Number : 7240005, Murcia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Hincelin-Mery A, Nicolas X, Cantalloube C, Pomponio R, Lewanczyk P, Benamor M, Ofengeim D, Krupka E, Hsiao-Nakamoto J, Eastenson A, Atassi N. Safety, pharmacokinetics, and target engagement of a brain penetrant RIPK1 inhibitor, SAR443820 (DNL788), in healthy adult participants. Clin Transl Sci. 2024 Jan;17(1):e13690. doi: 10.1111/cts.13690. Epub 2023 Dec 11. PMID 38010108

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 34 centers in 10 countries. A total of 190 participants were screened between 19 December 2022 and 15 September 2023, of which 16 were screen failures. Screen failures were due to not meeting the eligibility criteria.
Pre-assignment Details: The study consisted of a screening period (4 weeks before randomization), treatment period (a 48-week double-blind in Part A, an 48-week open-label in Part B, with a maximum total study duration of 100 weeks. A total of 174 participants were randomized and 173 were treated in the study. The study was terminated as it did not meet its primary and key secondary endpoints, therefore Week 96 data was not collected.
Groups:
- Part A: Placebo: Participants received placebo matching SAR443820 tablet orally once daily (QD) for 48 weeks in Part A.
- Part A: SAR443820: Participants received SAR443820 20 milligram (mg) tablet orally QD for 48 weeks in Part A.
- Part B: Placebo/SAR443820: Participants who had received placebo matching SAR443820 tablet in Part A, received SAR443820 20 mg tablet orally QD for 48 weeks during Part B.
- Part B: SAR443820/SAR443820: Participants who had received SAR443820 tablet in Part A, continued to receive SAR443820 20 mg tablet orally QD for 48 weeks during Part B.
Period: Part A (Double-blind Period: 48 Weeks)
Arm/Group | Part A: Placebo | Part A: SAR443820 | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Started | 86 | 88 | 0 | 0
Randomized and Treated | 86 | 87 | 0 | 0
Completed | 77 | 68 | 0 | 0
Not Completed | 9 | 20 | 0 | 0
Not completed — Other | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 3 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 13 | 0 | 0
Not completed — Randomized and not treated | 0 | 1 | 0 | 0
Period: Part B (Open-label Period: 48 Weeks)
Arm/Group | Part A: Placebo | Part A: SAR443820 | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Started | 0 | 0 | 77 | 68
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 77 | 68
Not completed — Study terminated by sponsor | 0 | 0 | 72 | 62
Not completed — Non-compliance with study schedule | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 3
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Randomized population=all participants from screened population who had been allocated to a randomized study treatment by interactive response technology (IRT) regardless of whether study treatment was received. Participants from Part A were allowed to transition to Part B per the study design hence baseline characteristics collected at the beginning of the study applies to both Part A and Part B.
Groups:
- Part A: Placebo: Participants received placebo matching SAR443820 tablet orally QD for 48 weeks in Part A.
- Part A: SAR443820: Participants received SAR443820 20 mg tablet orally QD for 48 weeks in Part A.
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: SAR443820 | Total
Number analyzed (Participants) | 86 | 88 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.27 (9.54) | 48.22 (8.21) | 47.75 (8.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 53 | 107
  Male | 32 | 35 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 69 | 74 | 143
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 11 | 20

OUTCOME MEASURES:

1. Secondary Outcome: Part A: Number of New Gadolinium-Enhancing T1 Hyperintense Lesions as Detected by Magnetic Resonance Imaging (MRI)
Description: The adjusted number of new Gd-enhancing T1 hyperintense lesions per scan were derived using negative binomial model.
Time Frame: Post-baseline (Baseline: Day 1, pre-dose) and up to Week 48
Population: Randomized and treated population consisted of all randomized participants who took at least 1 dose of study treatment.
Measure: Mean (95% Confidence Interval); unit: new Gd-enhancing T1 lesions per scan
Arm/Group | Part A: Placebo | Part A: SAR443820
Number analyzed (Participants) | 86 | 87
new Gd-enhancing T1 lesions per scan | 0.043 [0.020 to 0.088] | 0.155 [0.071 to 0.337]

2. Secondary Outcome: Part B: Number of New Gadolinium-Enhancing T1 Hyperintense Lesions as Detected by MRI
Description: Cumulative number of new Gd-enhancing T1 hyperintense lesions detected by MRI, defined as the sum of the individual number of new Gd-enhancing T1 hyperintense lesions at all scheduled visits calculated for each arm/group as a whole.
Time Frame: From Week 48 to approximately up to Week 72
Population: Randomized and treated population consisted of all randomized participants who took at least 1 dose of study treatment. Here, number of participants analyzed = participants with >=1 new enlarging T1-hyperintense lesions.
Measure: Number; unit: new Gd-enhancing T1 lesions
Arm/Group | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 5 | 4
new Gd-enhancing T1 lesions | 14 | 13

3. Secondary Outcome: Part A: Number of New, Enlarging T2 Hyperintense Lesions as Detected by MRI
Description: The adjusted number of new, enlarging T2 hyperintense lesions per year were derived using negative binomial model.
Time Frame: Post-baseline (Baseline: Day 1, pre-dose) and up to Week 48
Population: Randomized and treated population consisted of all randomized participants who took at least 1 dose of study treatment.
Measure: Mean (95% Confidence Interval); unit: new and enlarging T2 lesions per year
Arm/Group | Part A: Placebo | Part A: SAR443820
Number analyzed (Participants) | 86 | 87
new and enlarging T2 lesions per year | 1.285 [0.645 to 2.561] | 2.532 [1.183 to 5.422]

4. Secondary Outcome: Part B: Number of New, Enlarging T2 Hyperintense Lesions as Detected by MRI
Description: Cumulative number of new, enlarging T2 hyperintense lesions detected by MRI, defined as the sum of the individual number of new, enlarging T2 hyperintense lesions at all scheduled visits at all scheduled visits calculated for each arm/group as a whole.
Time Frame: From Week 48 to approximately up to Week 72
Population: Randomized and treated population consisted of all randomized participants who took at least 1 dose of study treatment. Here, number of participants analyzed = participants with >=1 new and/or enlarging T2-hyperintense lesions.
Measure: Number; unit: new and enlarging T2 lesions
Arm/Group | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 12 | 9
new and enlarging T2 lesions | 42 | 57

5. Secondary Outcome: Part A: Time to Onset of 12 Weeks Confirmed Disability Progression (CDP) From Baseline as Assessed by the Expanded Disability Status Scale (EDSS) Score
Description: Time to onset of 12 weeks CDP was defined as time from randomization to onset of an increase in EDSS score (defined as an increase of >=1.0 point from baseline EDSS score when baseline score was <=5.5 or an increase of >=0.5 points from baseline EDSS score when baseline score was >5.5) confirmed after a 12 weeks interval. EDSS was a scale for assessing neurologic impairment in participants with MS, based on 7 functional systems (FS) in brain which was used to derive score. The standard EDSS assessments of 7 FS (visual, brain stem, pyramidal, cerebellar, sensory, bowel/bladder, and cerebral functions) scoring was performed by assessment of neurologic symptoms in each FS. Ambulation scoring was done to conclude evaluation. Individual FS scores were then used in conjugation with ambulation score to obtain EDSS score which ranged from 0 (normal) to 10 (death due to MS), with higher scores indicating greater disability. Baseline was defined as Day 1 (pre-dose).
Time Frame: Baseline (Day 1, pre-dose) and Week 48
Population: Randomized and treated population consisted of all randomized participants who took at least 1 dose of study treatment. Only participants with data collected at baseline and Week 48 are reported.
Measure: Median (Full Range); unit: weeks
Arm/Group | Part A: Placebo | Part A: SAR443820
Number analyzed (Participants) | 6 | 6
weeks | 12.29 [11.9 to 24.3] | 24.14 [11.7 to 36.7]

6. Secondary Outcome: Part B: Time to Onset of 24 Weeks Confirmed Disability Progression From Baseline as Assessed by the Expanded Disability Status Scale Score
Description: Time to onset of 24 weeks CDP was defined as time from randomization to onset of an increase in EDSS score (defined as an increase of >=1.0 point from baseline EDSS score when baseline score was <=5.5 or an increase of >=0.5 points from baseline EDSS score when baseline score was >5.5) confirmed after a 12 weeks interval. EDSS was a scale for assessing neurologic impairment in participants with MS, based on 7 FS in brain which was used to derive score. The standard EDSS assessments of 7 FS (visual, brain stem, pyramidal, cerebellar, sensory, bowel/bladder, and cerebral functions) scoring was performed by assessment of neurologic symptoms in each FS. Ambulation scoring was done to conclude evaluation. Individual FS scores were then used in conjugation with ambulation score to obtain EDSS score which ranged from 0 (normal) to 10 (death due to MS), with higher scores indicating greater disability. Baseline was defined as Day 1 (pre-dose).
Time Frame: Baseline (Day 1, pre-dose) and approximately up to Week 72
Population: Randomized and treated population consisted of all randomized participants who took at least 1 dose of study treatment. Only participants with data collected at specified timepoints are reported.
Measure: Median (Full Range); unit: weeks
Arm/Group | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 5 | 3
weeks | 12.43 [12.1 to 24.3] | 24.14 [24.1 to 24.4]

7. Secondary Outcome: Part A: Time to Onset of Sustained 20% Increase in 9-Hole Peg Test (9-HPT) Confirmed Over at Least 12 Weeks
Description: The 9-HPT was a brief, standardized, quantitative test of upper extremity function (lower bound: 10 seconds; upper bound: 300 seconds). Two consecutive trials with the dominant hand were immediately followed by 2 consecutive trials with the non-dominant hand. The mean time to test completion served as an assessment of the participant's hand dexterity. A participant was asked to place pegs into holes and remove them with the dominant and non-dominant hand for several repetitions. A higher value of overall 9-HPT was indicative of higher disability. An increase of >=20% from the baseline score in the 9-HPT was considered meaningful worsening. Baseline was defined as Day 1 (pre-dose).
Time Frame: Baseline (Day 1, pre-dose) and Week 48
Population: as for outcome 5
Measure: Median (Full Range); unit: weeks
Arm/Group | Part A: Placebo | Part A: SAR443820
Number analyzed (Participants) | 3 | 3
weeks | 35.86 [11.9 to 36.1] | 12.14 [11.1 to 36.1]

8. Secondary Outcome: Part B: Time to Onset of Sustained 20% Increase in 9-Hole Peg Test Confirmed Over at Least 24 Weeks
Description: The 9-HPT was a brief, standardized, quantitative test of upper extremity function (lower bound: 10 seconds; upper bound: 300 seconds). Two consecutive trials with the dominant hand were immediately followed by 2 consecutive trials with the non-dominant hand. The mean time to test completion served as an assessment of the participant's hand dexterity. A participant was asked to place pegs into holes and remove them with the dominant and non-dominant hand for several repetitions. A higher value of overall 9-HPT was indicative of higher disability. An increase of >20% from the baseline score in the 9-HPT was considered meaningful worsening. Baseline was defined as Day 1 (pre-dose).
Time Frame: Baseline (Day 1, pre-dose) and approximately up to Week 72
Population: as for outcome 6
Measure: Median (Full Range); unit: weeks
Arm/Group | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 1 | 0
weeks | 36.1 [36.1 to 36.1] |

9. Secondary Outcome: Part A: Time to Onset of Sustained 20% Increase in Timed 25-Foot Walk Test (T25-FW) Confirmed Over at Least 12 Weeks
Description: The T25-FW test was used to assess a participant's walking ability, time in seconds to walk 25 feet (lower bound: 2.2 seconds; upper bound: 180 seconds). The participant was directed to 1 end of a clearly marked 25-foot course and was instructed to walk 25 feet as quickly as safely possible with several repetitions. The mean walk time was used for assessment of the participant's walking ability. An increase of >20% from the baseline score in the T25-FW test was considered as meaningful worsening. Baseline was defined as Day 1 (pre-dose).
Time Frame: Baseline (Day 1, pre-dose) and Week 48
Population: as for outcome 5
Measure: Median (Full Range); unit: weeks
Arm/Group | Part A: Placebo | Part A: SAR443820
Number analyzed (Participants) | 16 | 8
weeks | 12.29 [11.6 to 35.9] | 18.00 [11.7 to 36.1]

10. Secondary Outcome: Part B: Time to Onset of Sustained 20% Increase in Timed 25-Foot Walk Test Confirmed Over at Least 24 Weeks
Description: The T25-FW test was used to assess a participant's walking ability, time in seconds to walk 25 feet (lower bound: 2.2 seconds; upper bound: 180 seconds). The participant was directed to one end of a clearly marked 25-foot course and was instructed to walk 25 feet as quickly as safely possible with several repetitions. The mean walk time was used for assessment of the participant's walking ability. An increase of >20% from the baseline score in the T25-FW test was considered as meaningful worsening. Baseline was defined as Day 1 (pre-dose).
Time Frame: Baseline (Day 1, pre-dose) and approximately up to Week 72
Population: as for outcome 6
Measure: Median (Full Range); unit: weeks
Arm/Group | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 8 | 8
weeks | 12.14 [11.6 to 24.3] | 18.00 [11.7 to 48.1]

11. Secondary Outcome: Parts A and B: Change From Baseline in Expanded Disability Status Scale Score
Description: EDSS was a scale for assessing neurologic impairment in participants with MS, based on 7 FS in the brain which was used to derive the EDSS (score). The standard EDSS assessments of 7 FS (visual, brain stem, pyramidal, cerebellar, sensory, bowel/bladder, and cerebral functions) scoring was performed by assessment of neurologic symptoms in each FS. Ambulation scoring was done to conclude the evaluation. Individual FS scores were then used in conjugation with ambulation score to obtain EDSS score which ranged from 0 (normal) to 10 (death due to MS), with higher scores indicating greater disability. A negative change from baseline indicates improvement. Baseline was defined as Day 1 (pre-dose).
Time Frame: Baseline (Day 1, pre-dose) and Week 48 (Part A) and approximately up to Week 72 (Part B)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Placebo | Part A: SAR443820 | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 78 | 76 | 3 | 1
score on a scale | -0.013 (0.611) | -0.023 (0.676) | -0.167 (0.722) | -1.000 (NA) — Standard deviation (SD) cannot be calculated for a single participant.

12. Secondary Outcome: Part A: Annualized Relapse Rate (ARR) of Relapsing Remitting Multiple Sclerosis (RMS) Population
Description: Relapse was defined as the occurrence of acute, new neurological symptoms or worsening of previous neurological symptoms with an objective change on neurological examination attributable to MS. Symptoms were as follows: attributed to MS, last for >=24 hours, present at normal body temperature, and preceded by >=30 days of clinical stability (no previous MS relapse). The adjusted ARR was derived using negative binomial model with the total number of relapses per participant occurring in the observation period.
Time Frame: Up to Week 48
Population: Randomized and treated population consisted of all randomized participants who took at least 1 dose of study treatment. Only participants with RMS (RRMS plus relapsing SPMS) are reported.
Measure: Number (95% Confidence Interval); unit: relapses per participant-year
Arm/Group | Part A: Placebo | Part A: SAR443820
Number analyzed (Participants) | 41 | 42
relapses per participant-year | NA [NA to NA] — NA indicates that the number, lower and upper limit of 95% confidence interval (CI) were not estimable due to insufficient number of participants with events. | NA [NA to NA] — NA indicates that the number, lower and upper limit of 95% CI were not estimable due to insufficient number of participants with events.

13. Secondary Outcome: Part B: Annualized Relapse Rate of Relapsing Remitting Multiple Sclerosis Population
Description: Relapse was defined as the occurrence of acute, new neurological symptoms or worsening of previous neurological symptoms with an objective change on neurological examination attributable to MS. Symptoms were as follows: attributed to MS, last for >=24 hours, present at normal body temperature, and preceded by >=30 days of clinical stability (no previous MS relapse). The unadjusted ARR was the total number of relapses that occurred during the observation period divided by the total participant years in the study.
Time Frame: Approximately up to Week 72
Population: as for outcome 12
Measure: Number; unit: relapses per participant-year
Arm/Group | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 41 | 42
relapses per participant-year | 0.052 | 0.172

14. Secondary Outcome: Parts A and B: Percent Change From Baseline in Brain Volume Loss (BVL) as Detected by Brain Magnetic Resonance Imaging
Description: The basic MRI scan was performed at all sites and used to evaluate BVL. Imaging measure to detect degree of atrophy or decrease in whole brain, cortical and/or thalamic volume, which was diagnostic evidence of disease progression and played a key role in long-term disability. Baseline was defined as Day 1 (pre-dose).
Time Frame: Baseline (Day 1, pre-dose) and Week 48 (Part A) and approximately up to Week 72 (Part B)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part A: Placebo | Part A: SAR443820 | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 72 | 71 | 5 | 4
percent change | -0.177 (0.426) | -0.397 (0.462) | -0.502 (0.526) | -0.462 (0.869)

15. Secondary Outcome: Part A: Volume of Slowly Expanding Lesions (SELs)
Description: The basic MRI scan was performed at all sites and used to evaluate volume of SELs. SELs represent chronic active lesions in MS where there is ongoing, smoldering inflammation primarily driven by activated microglia and macrophages at the lesion edges. This localized, radial expansion causes gradual enlargement of pre-existing T2 MRI lesions over time and leads to progressive neural tissue damage including demyelination, axonal loss, and irreversible central nervous system (CNS) injury.
Time Frame: Week 48
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: microliter (µL)
Arm/Group | Part A: Placebo | Part A: SAR443820
Number analyzed (Participants) | 71 | 71
microliter (µL) | 5.436 [4.773 to 6.099] | 5.672 [4.958 to 6.386]

16. Secondary Outcome: Part B: Volume of Slowly Expanding Lesions
Description: The basic MRI scan was performed at all sites and used to evaluate volume of SELs. SELs represent chronic active lesions in MS where there is ongoing, smoldering inflammation primarily driven by activated microglia and macrophages at the lesion edges. This localized, radial expansion causes gradual enlargement of pre-existing T2 MRI lesions over time and leads to progressive neural tissue damage including demyelination, axonal loss, and irreversible CNS injury.
Time Frame: Approximately up to Week 72
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: µL
Arm/Group | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 5 | 4
µL | 1485.00 (2657.22) | 1152.00 (998.67)

17. Secondary Outcome: Part A: Number of Slowly Expanding Lesions
Description: The basic MRI scan was performed at all sites and used to evaluate number of SELs. SELs represent chronic active lesions in MS where there is ongoing, smoldering inflammation primarily driven by activated microglia and macrophages at the lesion edges. This localized, radial expansion causes gradual enlargement of pre-existing T2 MRI lesions over time and leads to progressive neural tissue damage including demyelination, axonal loss, and irreversible CNS injury.
Time Frame: Week 48
Population: Randomized and treated population consisted of all randomized participants who took at least 1 dose of study treatment. Participants were analyzed according to the intervention allocated by randomization. Only participants with data collected at specified timepoints are reported.
Measure: Least Squares Mean (95% Confidence Interval); unit: number of SEL
Arm/Group | Part A: Placebo | Part A: SAR443820
Number analyzed (Participants) | 71 | 71
number of SEL | 1.507 [1.296 to 1.718] | 1.534 [1.307 to 1.761]

18. Secondary Outcome: Part B: Number of Slowly Expanding Lesions
Description: as for outcome 17
Time Frame: Approximately up to Week 72
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: number of SEL
Arm/Group | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 5 | 4
number of SEL | 6.60 (9.84) | 6.25 (5.32)

19. Secondary Outcome: Part A: Normalized T1 Intensity of Slowly Expanding Lesions
Description: The basic MRI scan was performed at all sites and used to evaluate normalization of T1 intensity of SELs. It was used to quantify tissue damage within SELs of MS, reflecting neuro-axonal loss and demyelination and correlating with clinical progression.
Time Frame: Baseline (Day 1, pre-dose), Weeks 12, 24, 36, and 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part A: Placebo | Part A: SAR443820
Number analyzed (Participants) | 61 | 71
ratio
  Baseline (Day 1, pre-dose) | -0.055 (0.346) | 0.008 (0.354)
  Week 12: number analyzed (Participants) | 59 | 71
  Week 12 | -0.066 (0.369) | -0.026 (0.325)
  Week 24: number analyzed (Participants) | 61 | 70
  Week 24 | -0.096 (0.352) | -0.031 (0.341)
  Week 36: number analyzed (Participants) | 61 | 65
  Week 36 | -0.107 (0.355) | -0.053 (0.350)
  Week 48: number analyzed (Participants) | 60 | 64
  Week 48 | -0.123 (0.357) | -0.058 (0.370)

20. Secondary Outcome: Part B: Normalized T1 Intensity of Slowly Expanding Lesions
Description: The basic MRI scan was performed at all sites and used to evaluate normalized T1 intensity of SELs. It was used to quantify tissue damage within SELs of MS, reflecting neuro-axonal loss and demyelination and correlating with clinical progression.
Time Frame: Week 48 and Week 72
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 3 | 3
ratio
  Week 48 | -0.342 (0.118) | -0.083 (0.241)
  Week 72 | -0.507 (0.236) | -0.183 (0.201)

21. Secondary Outcome: Part A: Change From Baseline in the Number of Phase Rim Lesions (PRL) Conducted at 3 Tesla (3T) Capable Sites
Description: The basic MRI scan sequences were performed at all sites and used to evaluate number of PRL. Phase rim lesions were a subtype of MS lesion identified by a paramagnetic edge indicative chronic smoldering inflammation linked to chronic active lesions. Baseline was defined as Day 1 (pre-dose).
Time Frame: Baseline (Day 1, pre-dose) and Weeks 12, 24, 36, and 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: phase rim lesions
Arm/Group | Part A: Placebo | Part A: SAR443820
Number analyzed (Participants) | 40 | 38
phase rim lesions
  Week 12 | 0.05 (0.22) | 0.00 (0.00)
  Week 24: number analyzed (Participants) | 38 | 35
  Week 24 | 0.11 (0.65) | 0.00 (0.00)
  Week 36: number analyzed (Participants) | 38 | 32
  Week 36 | 0.11 (0.83) | 0.00 (0.00)
  Week 48: number analyzed (Participants) | 36 | 32
  Week 48 | 0.14 (1.02) | -0.03 (0.18)

22. Secondary Outcome: Part B: Change From Baseline in the Number of Phase Rim Lesions Conducted at 3 Tesla Capable Sites
Description: as for outcome 21
Time Frame: Baseline (Day 1, pre-dose) and approximately up to Week 72
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: phase rim lesions
Arm/Group | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 3 | 4
phase rim lesions | 2.33 (4.93) | -0.25 (0.50)

23. Secondary Outcome: Parts B and A+B: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs) After SAR443820 Initiation
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAEs were defined as the AEs that developed, worsened or became serious during the treatment-emergent period (defined as time from first administration of study treatment (Day 1) to last administration of study treatment + 14 days). SAE: Any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. All TEAE occurring after SAR443820 initiation are provided for both randomized treatment arms in this endpoint.
Time Frame: From first dose of SAR443820 (Day 1, post-dose) up to 14 days after last dose of SAR443820 administration in Part B, approximately 93 weeks for Parts A+B combined arm (SAR443820/SAR443820), approximately 45 weeks Part B Arm (Placebo/SAR443820)
Population: Safety population consisted of all randomized participants who took at least 1 dose of SAR443820. All participants from safety population and treated with SAR443820 are included in Part B arm and participants from safety population are included in Parts A+B arm. The combined safety analysis for TEAE provided the accurate summary of all TEAE in both treatment groups after the initiation of SAR443820.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Placebo/SAR443820: Participants who had received placebo matching SAR443820 tablet in Part A for 48 weeks, received first intake of SAR443820 20 mg tablet orally QD up to 48 weeks during Part B.
- Parts A+B: SAR443820/SAR443820: Participants who had received SAR443820 tablet in Part A for 48 weeks, continued to receive SAR443820 20 mg tablet orally QD up to 48 weeks during Part B.
Arm/Group | Part B: Placebo/SAR443820 | Parts A+B: SAR443820/SAR443820
Number analyzed (Participants) | 77 | 164
Participants
  TEAEs | 39 | 108
  TESAEs | 5 | 7

24. Secondary Outcome: Part A: Plasma Concentration of SAR443820
Description: Plasma samples were collected at specified timepoints to determine plasma concentrations of SAR443820.
Time Frame: Day 1: 0.25-1 hour and 1-3 hours post-dose; Week 2: pre-dose, 0.5-3 hours post-dose; Weeks 6, 12, and 36: pre-dose
Population: Pharmacokinetic (PK) population consisted of all randomized and treated participants with at least 1 post-baseline PK result with adequate documentation of dosing and sampling dates and times. Only participants who received SAR443820 with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: nanogram/mL
Units Other Than Participants: Samples
Groups:
- Part A: SAR443820: Participants received SAR443820 20 mg tablet orally QD for 48 weeks during Part A.
Arm/Group | Part A: SAR443820
Number analyzed (Participants) | 87
Number analyzed (Samples) | 540
nanogram/mL
  Day 1: 0.25-1 hours post-dose: number analyzed (Samples) | 79
  Day 1: 0.25-1 hours post-dose | 205.450 (134.734)
  Day 1: 1-3 hours post-dose: number analyzed (Samples) | 82
  Day 1: 1-3 hours post-dose | 237.232 (92.001)
  Week 2: pre-dose: number analyzed (Samples) | 81
  Week 2: pre-dose | 52.841 (54.432)
  Week 2: 0.5-3 hours post-dose: number analyzed (Samples) | 83
  Week 2: 0.5-3 hours post-dose | 289.312 (129.688)
  Week 6: pre-dose: number analyzed (Samples) | 83
  Week 6: pre-dose | 45.230 (41.458)
  Week 12: pre-dose: number analyzed (Samples) | 75
  Week 12: pre-dose | 49.039 (41.203)
  Week 36: pre-dose: number analyzed (Samples) | 57
  Week 36: pre-dose | 56.461 (60.180)

25. Secondary Outcome: Part B: Time to Onset of Composite Confirmed Disability Progression Confirmed Over at Least 24 Weeks
Description: Time to onset of 24-week CCDP, was assessed by composite endpoint EDSS-Plus (EDSS score, or T25-FW test, or 9-HPT), was confirmed over at least 24 week. The EDSS-plus event was defined as disability progression on at least 1 of 3 components, EDSS score, or T25-FW test, or 9-HPT. Disability criteria for the individual components are defined as follows: Disability progression on the EDSS was defined as an increase of >=1.0 point from the baseline EDSS score when the baseline score was <=5.5 or an increase of >=0.5 points from the baseline EDSS score when the baseline score was >5.5. Disability progression on the T25-FW test was defined as an increase (worsening) of >=20% from the baseline score. Disability progression on the 9-HPT was defined as an increase (worsening) of >=20% from the baseline score. Baseline was defined as Day 1 (pre-dose).
Time Frame: Baseline (Day 1, pre-dose) and approximately up to Week 72
Population: as for outcome 6
Measure: Median (Full Range); unit: weeks
Arm/Group | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 12 | 10
weeks | 12.29 [11.6 to 36.1] | 24.00 [11.7 to 48.1]

26. Secondary Outcome: Part B: Change From Baseline in Multiple Sclerosis Impact Scale-29 Version 2 (MSIS-29v2) Physical and Psychological Domains Scores
Description: The MSIS-29v2 evaluates the specific physical and psychological impact of MS from a participant's perspective. This participant reported outcome instrument has 2 subscales: a physical impact score (20 items) and a psychological impact score (9 items). The physical and psychological impact subscales of the MSIS-29v2 range from 0 to 100, with higher scores indicating greater physical or psychological impact. Each of the 2 scales are scored by summing the responses across items, then converting to score range 0-100 where 100 indicates greater impact of disease on daily function (worse health). Baseline was defined as Day 1 (pre-dose).
Time Frame: Baseline (Day 1, pre-dose) and approximately up to Week 72
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 4 | 3
score on a scale
  Physical domains score | 11.667 (28.447) | 2.222 (1.925)
  Psychological domains score | 13.889 (52.498) | 4.938 (5.658)

27. Secondary Outcome: Part B: Change From Baseline in Multiple Sclerosis Walking Scale 12 Items (MSWS-12) Scores
Description: The MSWS-12 measured the impact of walking impairment in participants with MS. This participant reported outcome instrument has 12 items with a global score ranging from 0 to 100. A higher score indicates better quality of life. The MSWS-12 score was calculated by summing the 12 components and transforming into a scale with a range of 0 to 100, with higher score indicating better quality of life. Baseline was defined as Day 1 (pre-dose).
Time Frame: Baseline (Day 1, pre-dose) and approximately up to Week 72
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 3 | 3
score on a scale | 4.861 (17.472) | -1.389 (6.365)

28. Primary Outcome: Part A: Change From Baseline to Week 48 in Serum Neurofilament Light Chain (sNfL) Levels
Description: Serum blood samples were collected at indicated time points to measure changes in NfL, a marker of neuronal damage. Baseline was defined as the average value of the assessments on screening and Day 1 visits prior to the first dose of the study treatment unless the number of Gadolinium (Gd)-enhancing T1 lesion at Day 1 was greater than zero in which case baseline was the lower value of screening and Day 1 visits.
Time Frame: Baseline (up to Day 1, pre-dose) and Week 48
Population: The modified intent-to-treat (mITT) population consisted of all randomized participants who took at least 1 dose of study treatment and with an evaluable primary endpoint. Only participants with data collected at baseline and Week 48 are reported.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Part A: Placebo | Part A: SAR443820
Number analyzed (Participants) | 80 | 85
picograms per milliliter (pg/mL)
  Baseline | 9.622 (5.316) | 10.319 (7.402)
  Week 48: number analyzed (Participants) | 74 | 68
  Week 48 | 0.958 (6.983) | -0.343 (7.761)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: SAR443820; Analysis was performed using mixed-effect model with repeated measures (MMRM) including the fixed categorical effects of the treatment group, multiple sclerosis (MS) clinical subtype (relapsing remitting multiple sclerosis [RRMS], secondary progressive multiple sclerosis [SPMS], or primary progressive multiple sclerosis [PPMS]), visit, treatment-by-visit interaction, log-transformed baseline sNfL levels and log-transformed baseline sNfL levels-by-visit interaction; Test type: Superiority; p = 0.8042, MMRM; LS Geometric Mean Ratio to Baseline = 0.986, 95% CI 2-sided [0.881 to 1.103]

29. Primary Outcome: Part B: Change From Baseline to Week 72 in Serum Neurofilament Light Chain Levels
Description: Serum blood samples were collected at indicated time points to measure changes in NfL, a marker of neuronal damage. Baseline was defined as the average value of the assessments on screening and Day 1 visits prior to the first dose of the study treatment unless the number of Gd-enhancing T1 lesion at Day 1 was greater than zero in which case baseline was the lower value of screening and Day 1 visits.
Time Frame: Baseline (up to Day 1, pre-dose) and Week 72
Population: The mITT population consisted of all randomized participants who took at least 1 dose of study treatment and with an evaluable primary endpoint. Only participants with data collected at baseline and Week 72 are reported.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
Number analyzed (Participants) | 80 | 85
pg/mL
  Baseline | 9.622 (5.316) | 10.319 (7.402)
  Week 72: number analyzed (Participants) | 28 | 25
  Week 72 | -0.320 (3.433) | -0.270 (5.247)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment (Day 1, post-dose) up to 14 days after last dose of study treatment administration, up to 50 weeks for Part A, and 45 weeks for Part B. All-cause mortality (death) was assessed from signing of the informed consent form (Week -4) to study termination, approximately 100 weeks.
Description: Analysis was performed on safety population.
Arm/Group | Part A: Placebo | Part A: SAR443820 | Part B: Placebo/SAR443820 | Part B: SAR443820/SAR443820
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/87 | 0/77 | 0/68
Serious Adverse Events (participants affected / at risk) | 1/86 | 2/87 | 5/77 | 0/68
Other Adverse Events (participants affected / at risk) | 37/86 | 43/87 | 15/77 | 8/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=86) | Part A: SAR443820 (N=87) | Part B: Placebo/SAR443820 (N=77) | Part B: SAR443820/SAR443820 (N=68)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple Sclerosis Relapse (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis Toxic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver Injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=86) | Part A: SAR443820 (N=87) | Part B: Placebo/SAR443820 (N=77) | Part B: SAR443820/SAR443820 (N=68)
Covid-19 (Infections and infestations) | 6 (6) | 8 (8) | 4 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (8) | 4 (4) | 1 (1) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (5) | 4 (4) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 4 (5) | 7 (8) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 6 (7) | 5 (7) | 3 (3) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (2) | 7 (8) | 3 (3) | 2 (3)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 6 (6) | 0 (0) | 2 (3)
Hepatic Enzyme Increased (Investigations) | 1 (1) | 15 (15) | 3 (3) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 9 (15) | 6 (8) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 7 (8) | 3 (4) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
The study was terminated as it did not meet its primary and key secondary endpoints, therefore Week 96 data was not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT05630547/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT05630547/SAP_001.pdf